CLINICAL TRIAL: NCT04600934
Title: Shockwave Assisted Large Bore Access (TAVR, TEVAR, EVAR, FEVAR)
Brief Title: Shockwave Assisted Large Bore Access
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Medical University of South Carolina (Other)
Collaborators: Shockwave Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Mathew Wooster, Assistant Professor, Medical University of South Carolina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00103170
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2023-09

CONDITIONS: Vascular Diseases
Keywords: Vascular Surgery
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard POBA (plain old balloon angioplasty) (Active Comparator): The first 50 patients will be pre-treated with standard POBA
  Interventions: Device: Plain old balloon angioplasty
- Shockwave (Experimental): The second 50 patients will be treated primarily with Shockwave
  Interventions: Device: Shockwave

INTERVENTIONS:
Device: Shockwave — Shockwave Medical, Inc. Peripheral Lithoplasty® System
  Arms: Shockwave
Device: Plain old balloon angioplasty — POBA
  Arms: Standard POBA (plain old balloon angioplasty)

SUMMARY:
Annually, 150-200 TAVR with unilateral large bore access and 200 combined TEVAR/EVAR/FEVAR with bilateral large bore access are performed at our institution. Nearly 50 percent of patients fall outside IFU for access vessel size. Adjuncts described include iliac conduit, crack and pave, balloon expandable sheaths, direct aortic puncture, transcaval delivery, alternative access point (i.e axillary, carotid). Each of these adjuncts comes with additional complication potential and by nature of being used less frequently than the standard femoral access makes the procedure more challenging.

The intervention the use of the Shockwave Medical, Inc. Peripheral Lithoplasty® System to achieve large bore access in patients whose vessels fall outside of the IFU suggested dimensions.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Indicated for planned procedure requiring large bore (>12 French sheath) access
* Mental capacity to provide informed consent
* Iliac access vessel demonstrates >50% circumferential calcium
* Iliac access vessel demonstrates maximum inner lumen diameter less than IFU for device required
* Iliac access vessel demonstrates maximum outer wall diameter greater than or equal to IFU for device required
* Preoperative CT angiogram, </= 5mm slices
* Preoperative ABI/TP
* Unsuccessful delivery of large bore sheath without adjunctive intervention

  o Definition of unsuccessful = operator assessment of the following
* Visible distortion of iliac artery calcification under fluoroscopy without forward progress of device
* Adverse forward pressure application by operator
* Failure of device to track with external pressure applied to abdomen
* Patient intolerance of advancement (pain response) in awake patient

Exclusion Criteria:

* Contraindicated for antiplatelet therapy (aspirin or plavix)
* Planned iliofemoral surgical reconstruction in next 30 days
* Prior common or external iliac artery stent placement
* Prior aorto-iliac, aorto-femoral, or iliofemoral bypass present
* Iliac access vessel demonstrates maximum outer wall diameter less than IFU for device required
* Inability to obtain preoperative CTA (contrast allergy, CKD, etc)
* Inability to traverse iliac segment with wire
* Emergent procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Successful advancement of planned large bore access device | Day 1
  Technical success-defined as successful advancement of planned large bore access device without use of additional adjuncts (stenting, repeat shockwave treatment, high pressure balloon, alternative access pathway)

CONTACTS AND LOCATIONS:
Overall Officials: Mathew Wooster, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States